CLINICAL TRIAL: NCT04484051
Title: Growth Hormone Study in Adults With Prader-Willi Syndroom
Brief Title: Growth Hormone Study in Adults With Prader-Willi Syndrome
Acronym: GAP
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Foundation for Prader-Willi Research (Other); Prader-Willi Fonds (Unknown)
Responsible Party: Principal Investigator, dr. Laura C. G. de Graaff-Herder, MD, PhD, Erasmus Medical Center
Other Study IDs: GAP
Record Dates: First submitted 2020-07-15; First posted 2020-07-23 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Growth hormone; Body composition; Cardiovascular disease
MeSH Terms: conditions — Prader-Willi Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Routine clinical care with Genotropin treatment: Data collection throughout routine clinical care with subcutaneous injections Genotropin, 0.6-0.8 mg/day. Participants start with 0.2 mg/day and the dose increases with 0.2 mg/day per month to a maximum dose of 0.6-0.8 mg/day.

SUMMARY:
The overall objective of this study is to measure the effect of growth hormone (GH) treatment on physical and psychosocial health in adults with Prader-Willi syndrome. Adults with PWS who have not been treated with GH during the past three years and who will start with GH treatment as part of regular patient care will be asked for informed consent to participate in this open-label prospective cohort study. We hypothesize that growth hormone treatment will improve the physical and psychosocial health.

DETAILED DESCRIPTION:
OBJECTIVES:

To measure the effect of GHt on physical and psychosocial health in adults with PWS.

The primary endpoint is change in lean body mass (LBM (kg)) as assessed by Dual Energy X-ray Absorptiometry (DEXA) scan. Secondary endpoints are total fat mass, bone density, physical health and psychosocial health. Also the occurrence of side-effects will be assessed. Only data that are collected as part of regular patient care will be used.

STUDY DESIGN:

Open-label prospective cohort study.

STUDY POPULATION:

Adults with PWS who have not been treated with GH during the past three years and who will start with GHt as part of regular patient care.

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed with Prader-Willi syndrome (genetically confirmed)

Exclusion Criteria:

* Non cooperative behaviour
* Pregnancy
* Known malignancies
* Poorly controlled diabetes (HbA1c > 64 mmol/mol (8%))
* Untreated obstructive sleep apnea (apnea-hypopnea index > 5)
* Body mass index above 40 kg/m2
* Upper-airway obstruction of any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with PWS who have not been treated with GH during the past three years and who will start with GHt as part of regular patient care.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-24 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in lean body mass | 36 months
  Change in lean body mass (in kg) as measured by Dual Energy X-ray Absorptiometry scan

SECONDARY OUTCOMES:
Change in fat mass | 36 months
  Change in fat mass (in kg) as measured by Dual Energy X-ray Absorptiometry scan
Change in bone density | 36 months
  Change in bone density (in T-score) as measured by Dual Energy X-ray Absorptiometry scan
Change in physical strength | 36 months
  Change in physical strenght as measured by handgrip dynamometer and sit-to-stand tests
Change in laboratory measurements | 36 months
  Changes in the following laboratory measurements:
  * Glycosylated hemoglobin (mmol/mol)
  * Total cholesterol (mmol/L)
  * Low-density lipoprotein cholesterol (mmol/L)
  * High-density lipoprotein cholesterol (mmol/L)
  * Insulin-like growth factor 1 (nmol/L)
  * Free thyroxine 4 (pmol/L)
  * Luteinizing hormone (U/I)
  * Follicle stimulating hormone (U/I)
  * Estradiol or testosterone (nmol/L)
  * Sex hormone binding globulin (nmol/L)
  * Aspartate transaminase (U/L)
  * Alanine transaminase (U/L)
  * Alkaline phosphatase (U/L)
  * Gamma glutamyl transpeptidase (U/L)
  * Total bilirubin (micromol/L)
  * Lactate dehydrogenase (U/L)
  * Urea (mmol/L)
  * Creatinine (micromol/L)
  * Hemoglobin (mmol/L)
  * Hematocrit (L/L)
  * Mean corpuscular volume (fL)
  * Leukocytes (10^9/L)
  * Thrombocytes (10^9/L)
  * 25-OH vitamin D (nmol/L)
Change in psychosocial functioning | 36 months
  Change in psychosocial functioning as estimated with the Adult Behaviour Checklist
Change in caregiver burden | 36 months
  Change in caregiver burden as estimated with the Zarit Burden Interview

OTHER OUTCOMES:
Change in weight and waist-hip ratio | 36 months
  Change in weight (in kg) and waist-hip ratio
Change in blood pressure | 36 months
  Change in blood pressure (in mmHg)
Occurence of side-effects | 36 months
  Occurrence of side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Laura de Graaff, MD, PhD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam
Locations (1):
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data has not been finalized yet. The investigators intent to share the full anonymized dataset, study protocol and statistical analysis plan upon request after publication of the results. Informed consent forms will not be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available around begin 2027 (after publication of the results). The data will be available for 15 years.
Access Criteria: Upon reasonable request.